CLINICAL TRIAL: NCT02602028
Title: The Comparison of the Efficacy of Once and Twice Daily Colchicine Dosage in Pediatric Patients With Familial Mediterranean Fever: A Randomized Trial
Brief Title: The Comparison of the Efficacy of Once and Twice Daily Colchicine Dosage in Pediatric Patients With FMF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Erkan Demirkaya, MD, MSc, Assoc. Prof., Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1491-1437-11/1539
Record Dates: First submitted 2015-11-05; First posted 2015-11-11 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Familial Mediterranean Fever
Keywords: Familial Mediterranean Fever; Colchicine
MeSH Terms: conditions — Familial Mediterranean Fever | interventions — Colchicine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- once daily dosage schema of colchicine (Experimental): The once daily dosage group was prescribed as once daily at 08:00 a.m. (Total 1mg)
  Interventions: Drug: colchicine
- twice daily dosage schema of colchicine (Experimental): Twice daily dosage group received the treatment twice daily at 08:00 a.m. and 08:00 p.m. (Total 1mg)
  Interventions: Drug: colchicine

INTERVENTIONS:
Drug: colchicine — to compare once daily dosage schema of colchicine and twice daily dosage schema of colchicine
  Other Names: colchicum

SUMMARY:
It was aimed to examine the efficacy and safety of once daily dosage schema of colchicine in pediatric patients with FMF compared to twice daily dosage schema.

In this 24-week, multicentric, randomized, controlled, noninferiority trial, pediatric patients newly diagnosed with FMF, carrying homozygote or compound heterozygote mutation and did not receive any treatment, were included. Patients were randomly assigned using block randomization method to receive treatment with once or twice daily doses. Clinical and laboratory characteristics and medication side effects were recorded and compared between groups. The study complied with Good Clinical Practice and the Consolidated Standards for Reporting of Trials (CONSORT) statement.

DETAILED DESCRIPTION:
Study design This study was conducted by members of the FMF Arthritis Vasculitis and Orphan disease Research in Pediatric Rheumatology (FAVOR, www.favor.org.tr) at 10 centers in Turkey. This is a multicentric randomized controlled, noninferiority trial of two parallel groups being followed up in pediatric rheumatology outpatient clinics. The randomization was done at baseline visit and patients were assessed in two more visits, three months apart. The study complied with Good Clinical Practice (GCP) and the Consolidated Standards for Reporting of Trials (CONSORT) statement.

Participants Inclusion criteria Pediatric patients who were newly diagnosed with Familial Mediterranean Fever according to Yalcinkaya or Tel-Hashomer criteria and who were confirmed with the genetic analysis as having compound heterozygote or homozygote mutation were enrolled. Eligible patients between ages of 5-16 and weighted 15-30 kg who and had not received any treatment were included. All patients included were asked the physicians to be proved and recorded as having at least one FMF attack before enrollment for the study.

Exclusion criteria Patients with a major congenital malformation, with a risk of pregnancy, and with other chronic diseases such as organ transplantation, hepatic disorder chronic kidney disease and AA amyloidosis, thyroid disease or rheumatologic disorders other than FMF, were excluded.

Baseline assessment and Outcome Measures At the baseline visit, medical history and complaints about the disease were questioned and physical examination and laboratory tests were performed. In following visits, any attack or findings due to colchicine since the last visit were investigated in addition to baseline visit.

Interventions The once daily dosage group was prescribed as once daily at 08:00 a.m. and the twice daily dosage group received the treatment twice daily at 08:00 a.m. and 08:00 p.m. Disease severity was assessed via Mor scoring system, modified for pediatric patients in all visits. A physician from each center was chosen to be responsible for data collection. After each visit the data was registered to a web-based registry system in "www.favor.org.tr" web site. To ensure accurate, complete, and reliable data, the following procedures were followed: data collection, encoding, and storage had been provided for the centers; a training session had been held to provide instruction on the protocol; periodic meetings had been held with study coordinators the principal investigator stayed in contact with the study coordinators by mail, telephone, and/or fax; and finally a data manager reviewed and evaluated the data.

Colchicine dosage The required colchicine dosage was calculated as total 1 mg daily according to internationally accepted advisory. All patients were prescribed 0.5 mg Colchicine tablets. Patients in once daily dosage group were given 2 tablets of Colchicine at 08.00 a.m. Twice daily dosage group received 1 tablet of 0,5 mg Colchicine at 08:00 a.m. and 1 tablet of 0,5 mg Colchicine at 08:00 p.m.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Familial Mediterranean Fever according to Yalcinkaya or
* Tel-Hashomer criteria
* Diagnosis confirmed with the genetic analysis as compound heterozygote or
* homozygote mutation
* Patients between ages of 5-16 and weighted 15-30 kg
* Not received any treatment for FMF

Exclusion criteria:

* Major congenital malformation
* Organ transplantation
* Hepatic disorder
* Chronic kidney disease
* AA amyloidosis
* Thyroid disease
* Rheumatologic disorders other than FMF

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 79 (Actual)
Dates: Start 2011-04; Primary Completion 2013-04 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Mor severity scoring system | At baseline and every 12 weeks, up to 24 weeks. Change in disease severity as assessed by the Mor severity scoring system.
  The primary objectives of this study were to compare the effectiveness of once and twice daily colchicine dosage regimens regarding taking control of disease symptoms which can be reducing disease severity which was assessed by modified Mor scoring system and
Adverse events | up to 24 weeks
  Adverse Events That Are Related to Treatment

SECONDARY OUTCOMES:
Number of Participants With Abnormal Laboratory Values | At baseline and every 12 weeks, up to 24 weeks.
  Laboratory findings such as erythrocyte sedimentation rate (ESR), C-reactive protein (CRP), serum amyloid A (SAA) levels were used for the indication of inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Erkan Demirkaya, MD, MSc, Principal Investigator — Saglik Bilimleri Universitesi Gulhane Tip Fakultesi; Cengizhan Acikel, MD, MPH, Study Chair — Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Locations (1):
- FMF Arthritis Vasculitis and Orphan Disease Research in Paediatric Rheumatology (FAVOR), Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Polat A, Acikel C, Sozeri B, Dursun I, Kasapcopur O, Gulez N, Simsek D, Saldir M, Dokurel I, Poyrazoglu H, Bakkaloglu S, Delibas A, Ekinci Z, Ayaz NA, Kandur Y, Peru H, Kurt YG, Polat SR, Unsal E, Makay B, Gok F, Ozen S, Demirkaya E; FMF Arthritis Vasculitis and Orphan Disease Research in Pediatric Rheumatology (FAVOR). Comparison of the efficacy of once- and twice-daily colchicine dosage in pediatric patients with familial Mediterranean fever--a randomized controlled noninferiority trial. Arthritis Res Ther. 2016 Apr 7;18:85. doi: 10.1186/s13075-016-0980-7. PMID 27055417